CLINICAL TRIAL: NCT01518101
Title: A Randomized, Open-label, Cross-over Study to Evaluate Patient Preferences for Eucreas® Versus Victoza® as add-on to Metformin in Type 2 Diabetes Mellitus Patients Who Did Not Have Adequate Glycaemic Control With Metformin.
Brief Title: Vildagliptin Versus Liraglutide - Patient Preference After Receiving Both Medications
Acronym: PREFER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLMF237ADE03; 2011-003818-16 (EudraCT Number)
Record Dates: First submitted 2012-01-22; First posted 2012-01-25 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes
Keywords: patient preference; vildagliptin; liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Preference | interventions — Vildagliptin; Metformin; Liraglutide

ARMS (2):
- Vildagliptin/Metformin followed by Liraglutide+Metformin (Experimental): In period I, Patients receiving vildagliptin will receive a stable dose of 50mg vildagliptin bid (twice daily) + 1000mg metformin bid for 12 weeks. In period II, patients will receive 0.6mg liraglutide od (once daily) + 1000mg metformin bid for the first week (week 13 - week 14) and increase the dose after 7 days up to 1.2mg liraglutide od/1000mg metformin bid.
  Interventions: Drug: Vildagliptin/ Metformin; Drug: Liraglutide; Drug: Metformin
- Liraglutide + Metformin followed by Vildagliptin/Metformin (Experimental): In period I, patients will receive 0.6mg liraglutide od (once daily) + 1000mg metformin bid (twice daily) for the first week (week 0 - week 1) and increase the dose after 7 days up to 1.2mg liraglutide od/1000mg metformin bid (week 2 -12). In period II, patients will receive a stable dose of 50mg vildagliptin bid (twice daily) + 1000mg metformin bid for next 12 weeks.
  Interventions: Drug: Vildagliptin/ Metformin; Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: Vildagliptin/ Metformin — Single pill combination of Vildagliptin/ Metformin (50/1000 mg).
Drug: Liraglutide — 1.2 mg once daily by commercially available injection pens
Drug: Metformin — 1000 mg tablets twice daily

SUMMARY:
Dipeptidyl peptidase-4 (DPP-4) inhibitors and glucagonlike peptide-1 (GLP-1) mimetics or analogs, which rely on the gastrointestinal hormones that are part of the incretin system for the treatment of T2DM, provide a therapeutic alternative to common oral antihyperglycemic agents (eg, sulfonylureas, thiazolidinediones). Although GLP-1 analogs and DPP-4 inhibitor medications are effective, there are differences between these products, including method of administration (injectable versus oral). Previous studies have shown that patients prefer additional oral agents over injectable agents because of fear of injections and the desire to avoid them. Patient preference is both clinically and financially important, as it can have long-term implications in terms of patients' motivation and insight into their disease state and its treatment, which might have a direct impact on the patient's compliance and treatment adherence. The aim of the current study is to evaluate the proportion of T2DM patients preferring oral anti-diabetic treatment with vildagliptin + metformin versus an injectable anti-diabetic treatment with liraglutide after 4 weeks of treatment with each medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Metformin monotherapy > 12 weeks
* Hemoglobin A1c (HbA1c) > 6.5 % and < 9.0 %
* Body mass Index (BMI) 19-35 (kg/m²)

Exclusion Criteria:

* acute diseases at randomization
* kidney diseases with creatinin > 120 µmol/l, glomerular filtration rate (GFR) <50 ml/min
* contraindication for Gliptins or glucagon-like-peptide-analogues according to the respective Summary of Product Characteristics (SmPC)
* previous use of dipeptidyl peptidase-4-inhibitors and GLP-1-mimetics

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients preferring each treatment regimen | At week 24
  Individual patient preference will be assessed by a two-choice question.

SECONDARY OUTCOMES:
Number of patients with treatment satisfaction for each treatment measured by Diabetes Treatment Satisfaction Questionnaire (TSQM-9) | week 12, Week 24
  The TSQM -9 is a psychometrically measure of the major dimensions of patients' satisfaction with medication. It provides scores on 3 scales: effectiveness (3 items), convenience (3 items) and global satisfaction (3 items).
Number of patients responding to subjective reasons of preference to each treatment | Week 12, week 24
  Individual patient preference will be assessed by a two-choice question. Patients will also be asked to specify the reason for preference. A specific questionnaire for the preference reasons will be provided.
Number of patients with adverse event, serious adverse events and death | 24 weeks
  Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Change from baseline in fasting plasma glucose at 12 weeks and 24 weeks | From Baseline to 12 weeks and 24 weeks
  Blood glucose measurements will be performed at baseline, week 12 and week 24 visits.
Change From Baseline in Hemoglobin A1c (HbA1c) at week 12 and week 24 | From Baseline to 12 weeks and 24 weeks
  HbA1c measurements will be performed at baseline, week 12 and week 24 visits.
Investigator preference and subjective reasons of preference to each treatment | Week 12, week 24
  Investigator preference will be assessed by a two-choice question. Investigator will also be asked to specify the reason for preference. A specific questionnaire for the preference reasons will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Germany (7):
  - Novartis Investigative Site, Völlkingen, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Meissen
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Saarlouis

REFERENCES:
- [Result] Ludemann J, Dutting ED, Dworak M. Patient preference and tolerability of a DPP-4 inhibitor versus a GLP-1 analog in patients with type 2 diabetes mellitus inadequately controlled with metformin: a 24-week, randomized, multicenter, crossover study. Ther Adv Endocrinol Metab. 2015 Aug;6(4):141-8. doi: 10.1177/2042018815595584. PMID 26301063